CLINICAL TRIAL: NCT04180267
Title: Efficacy of Low-magnitude High-frequency Vibration (LMHFV) on Musculoskeletal Health of Subjects on Wheelchair, a Randomized Controlled Study.
Brief Title: RCT of Vibration Effect on Vertebral BMD in Disabled Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinued due to COVID, community centres unable to provide services
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: V-Health Limited (Unknown)
Responsible Party: Principal Investigator, Professor CHEUNG Wing hoi, Louis, Associate Professor of Orthopaedics and Traumatology, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CREC 2019.087
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Vibration Therapy; Wheelchair; Osteoporosis
Keywords: Osteoporosis; Vibration Therapy; Disabled patient; Vertebral BMD
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: Subject will be randomized to either LMHFV group or control group. Subject assigned to LMHFV group will receive Low-magnitude High-frequency Vibration (35Hz, 0.3g, 20min/day, at least 3 times/week) for half year. The primary outcome is the effect of LMHFV on BMD at the lumbar spine, it will be assessed by dual-energy X-ray absorptiometry (DXA) that is clinically recommended for the diagnosis of osteoporosis. Secondary outcomes include muscle strength assessment, balancing ability and quality of life (QoL). All primary and secondary outcome assessments for all groups will be performed in the investigators' institute at baseline and 6 months post treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Subject assigned to Control Group will not receive LMHFV
- LMHFV group (Active Comparator): Subject assigned to LMHFV group will receive LMHFV (35Hz, 0.3g, 20min/day, at least 3 times/week) for half year.
  Interventions: Device: Low-magnitude High-frequency Vibration

INTERVENTIONS:
Device: Low-magnitude High-frequency Vibration — 35Hz, 0.3g, 20min/day, at least 3 times/week
  Other Names: Vibration Treatment
  Arms: LMHFV group

SUMMARY:
Osteoporosis is an age-related disease with progressive loss of bone, leading to fragile bone. It is one of the major health issues in elderly and causes medical, social and economic impacts globally. Patients with osteoporosis have high risk of osteoporotic fractures. Low-magnitude high-frequency vibration (LMHFV) is a non-invasive biophysical intervention providing whole-body mechanical stimulation. Previous studies showed that LMHFV is beneficial to muscle strength(1), postural control(2), balancing ability(3, 4), new bone formation(5-7), spinal bone mineral density (BMD)(8), and blood circulation(9). During the LMHFV treatment, elderly needs to stand upright on the platform for 20min/day. However, some elderlies with poor standing ability cannot stand for a long period. Therefore, the design of vibration platform is modified for the disabled patients and the efficacy of LMHFV on this group of elderlies will be verified. It is hypothesized that new design of LMHFV is beneficial to wheelchair users in terms of vertebral bone mineral density, muscle health and musculoskeletal functions.

DETAILED DESCRIPTION:
This study is a single-blinded randomized controlled trial to investigate the effect of LMHFV on vertebral BMD, muscle health, balancing ability and functional ability in wheelchair users (mainly on wheelchair for outdoor activities).

Healthy elderlies aged 65 years or above, with walking difficulties and using wheelchair are eligible. We exclude anyone who: [1] cannot stand and walk independently, [2] have vibration treatment before, [3] with malignancy, [4] with acute fractures or severe osteoarthritis (18), [5] with cardiovascular concern such as with pace-maker in-situ, [6] with chronic inflammatory conditions known to affect muscle metabolism such as rheumatoid arthritis, and [7] with high frequency of physical activities, such as subjects who participated in regular exercise five times a week or more.

Recruited subjects will be randomized to either LMHFV or control group. Subject assigned to LMHFV group will receive LMHFV (35Hz, 0.3g, 20min/day, at least 3 times/week) for 6 months. The primary outcome is BMD at the lumbar spine to be assessed by dual-energy X-ray absorptiometry (DXA) that is clinically recommended for the diagnosis of osteoporosis. All primary and secondary outcome assessments for all groups will be performed in the investigators' institute at baseline and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both genders aged ≥ 65 years
2. Wheelchair users with walking difficulties
3. Subjects with good general health conditions

Exclusion Criteria:

1. Subjects cannot stand and walk independently
2. Subjects who had vibration treatment before
3. Subjects with malignancy
4. Subjects with acute fractures or severe osteoarthritis
5. Subjects with cardiovascular concern such as with pace-maker in-situ
6. Subjects with chronic inflammatory conditions known to affect muscle metabolism such as rheumatoid arthritis
7. Subjects with high frequency of physical activities, such as subjects who participated in regular exercise five times a week or more

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Vertebral BMD | Half year
  BMD will be assessed by standard DXA equipment (Delphi W, Hologic, Waltham, MA, USA) which is a gold standard assessment for osteoporosis recommended by World Health Organization (WHO). Spine and hip are the two sites used for the diagnosis of osteoporosis and will be both performed.

SECONDARY OUTCOMES:
Muscle strength assessment | Half year
  Handgrip strength and quadriceps strength
Modified functional reach test | Half year
  Fall risk assessment for dynamic sitting balance
Biodex Balance System | Half year
  Postural stability test
36-item Short-Form Health Survey (SF-36) | Half year
  Assessment of health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Wing-hoi CHEUNG, Prof, Principal Investigator — CUHK
Locations (3):
- Hong Kong (3):
  - ELCHK, Shan King Care And Attention Home For The Elderly, Hong Kong
  - Evangelical Lutheran Church Social Service - Hong Kong, Hong Kong
  - Sun Chui Lutheran Centre For The Elderly, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torvinen S, Kannus P, Sievanen H, Jarvinen TA, Pasanen M, Kontulainen S, Nenonen A, Jarvinen TL, Paakkala T, Jarvinen M, Vuori I. Effect of 8-month vertical whole body vibration on bone, muscle performance, and body balance: a randomized controlled study. J Bone Miner Res. 2003 May;18(5):876-84. doi: 10.1359/jbmr.2003.18.5.876. PMID 12733727
- [Background] Rubin C, Recker R, Cullen D, Ryaby J, McCabe J, McLeod K. Prevention of postmenopausal bone loss by a low-magnitude, high-frequency mechanical stimuli: a clinical trial assessing compliance, efficacy, and safety. J Bone Miner Res. 2004 Mar;19(3):343-51. doi: 10.1359/JBMR.0301251. Epub 2003 Dec 22. PMID 15040821
- [Background] Verschueren SM, Roelants M, Delecluse C, Swinnen S, Vanderschueren D, Boonen S. Effect of 6-month whole body vibration training on hip density, muscle strength, and postural control in postmenopausal women: a randomized controlled pilot study. J Bone Miner Res. 2004 Mar;19(3):352-9. doi: 10.1359/JBMR.0301245. Epub 2003 Dec 22. PMID 15040822
- [Background] Stewart JM, Karman C, Montgomery LD, McLeod KJ. Plantar vibration improves leg fluid flow in perimenopausal women. Am J Physiol Regul Integr Comp Physiol. 2005 Mar;288(3):R623-9. doi: 10.1152/ajpregu.00513.2004. Epub 2004 Oct 7. PMID 15472009
- [Background] Mithal A, Bansal B, Kyer CS, Ebeling P. The Asia-Pacific Regional Audit-Epidemiology, Costs, and Burden of Osteoporosis in India 2013: A report of International Osteoporosis Foundation. Indian J Endocrinol Metab. 2014 Jul;18(4):449-54. doi: 10.4103/2230-8210.137485. No abstract available. PMID 25143898
- [Background] Morse LR, Nguyen N, Battaglino RA, Guarino AJ, Gagnon DR, Zafonte R, Garshick E. Wheelchair use and lipophilic statin medications may influence bone loss in chronic spinal cord injury: findings from the FRASCI-bone loss study. Osteoporos Int. 2016 Dec;27(12):3503-3511. doi: 10.1007/s00198-016-3678-4. Epub 2016 Jul 13. PMID 27412619
- [Background] Paleg G, Livingstone R. Systematic review and clinical recommendations for dosage of supported home-based standing programs for adults with stroke, spinal cord injury and other neurological conditions. BMC Musculoskelet Disord. 2015 Nov 17;16:358. doi: 10.1186/s12891-015-0813-x. PMID 26576548
- [Background] Menendez H, Ferrero C, Martin-Hernandez J, Figueroa A, Marin PJ, Herrero AJ. Acute effects of simultaneous electromyostimulation and vibration on leg blood flow in spinal cord injury. Spinal Cord. 2016 May;54(5):383-9. doi: 10.1038/sc.2015.181. Epub 2015 Oct 13. PMID 26458973
- [Background] Gao KL, Chan KM, Purves S, Tsang WWN. Reliability of dynamic sitting balance tests and their correlations with functional mobility for wheelchair users with chronic spinal cord injury. J Orthop Translat. 2014 Aug 7;3(1):44-49. doi: 10.1016/j.jot.2014.07.003. eCollection 2015 Jan. PMID 30035039
- [Background] Williams B, Allen B, Hu Z, True H, Cho J, Harris A, Fell N, Sartipi M. Real-Time Fall Risk Assessment Using Functional Reach Test. Int J Telemed Appl. 2017;2017:2042974. doi: 10.1155/2017/2042974. Epub 2017 Jan 10. PMID 28167961
- [Background] Ruhe A, Fejer R, Walker B. Center of pressure excursion as a measure of balance performance in patients with non-specific low back pain compared to healthy controls: a systematic review of the literature. Eur Spine J. 2011 Mar;20(3):358-68. doi: 10.1007/s00586-010-1543-2. Epub 2010 Aug 19. PMID 20721676
- [Background] Lam CL, Gandek B, Ren XS, Chan MS. Tests of scaling assumptions and construct validity of the Chinese (HK) version of the SF-36 Health Survey. J Clin Epidemiol. 1998 Nov;51(11):1139-47. doi: 10.1016/s0895-4356(98)00105-x. PMID 9817131
- [Result] Roelants M, Delecluse C, Verschueren SM. Whole-body-vibration training increases knee-extension strength and speed of movement in older women. J Am Geriatr Soc. 2004 Jun;52(6):901-8. doi: 10.1111/j.1532-5415.2004.52256.x. PMID 15161453
- [Result] Rogan S, Hilfiker R, Herren K, Radlinger L, de Bruin ED. Effects of whole-body vibration on postural control in elderly: a systematic review and meta-analysis. BMC Geriatr. 2011 Nov 3;11:72. doi: 10.1186/1471-2318-11-72. PMID 22054046
- [Result] Cheung WH, Mok HW, Qin L, Sze PC, Lee KM, Leung KS. High-frequency whole-body vibration improves balancing ability in elderly women. Arch Phys Med Rehabil. 2007 Jul;88(7):852-7. doi: 10.1016/j.apmr.2007.03.028. PMID 17601464
- [Result] Leung KS, Li CY, Tse YK, Choy TK, Leung PC, Hung VW, Chan SY, Leung AH, Cheung WH. Effects of 18-month low-magnitude high-frequency vibration on fall rate and fracture risks in 710 community elderly--a cluster-randomized controlled trial. Osteoporos Int. 2014 Jun;25(6):1785-95. doi: 10.1007/s00198-014-2693-6. Epub 2014 Mar 28. PMID 24676848
- [Result] Chung SL, Leung KS, Cheung WH. Low-magnitude high-frequency vibration enhances gene expression related to callus formation, mineralization and remodeling during osteoporotic fracture healing in rats. J Orthop Res. 2014 Dec;32(12):1572-9. doi: 10.1002/jor.22715. Epub 2014 Aug 17. PMID 25131218
- [Result] Wang J, Leung KS, Chow SK, Cheung WH. The effect of whole body vibration on fracture healing - a systematic review. Eur Cell Mater. 2017 Sep 7;34:108-127. doi: 10.22203/eCM.v034a08. PMID 28880360
- [Result] Choi SJ, Shin WS, Oh BK, Shim JK, Bang DH. Effect of training with whole body vibration on the sitting balance of stroke patients. J Phys Ther Sci. 2014 Sep;26(9):1411-4. doi: 10.1589/jpts.26.1411. Epub 2014 Sep 17. PMID 25276025
- [Result] Zhu TY, Hung VW, Cheung WH, Cheng JC, Qin L, Leung KS. Value of Measuring Bone Microarchitecture in Fracture Discrimination in Older Women with Recent Hip Fracture: A Case-control Study with HR-pQCT. Sci Rep. 2016 Sep 27;6:34185. doi: 10.1038/srep34185. PMID 27670149
- [Result] Cheung WH, Li CY, Zhu TY, Leung KS. Improvement in muscle performance after one-year cessation of low-magnitude high-frequency vibration in community elderly. J Musculoskelet Neuronal Interact. 2016 Mar;16(1):4-11. PMID 26944817
- [Derived] Chow SKH, Ho CY, Wong HW, Chim YN, Wong RMY, Cheung WH. Efficacy of low-magnitude high-frequency vibration (LMHFV) on musculoskeletal health of participants on wheelchair: a study protocol for a single-blinded randomised controlled study. BMJ Open. 2020 Dec 15;10(12):e038578. doi: 10.1136/bmjopen-2020-038578. PMID 33323430